CLINICAL TRIAL: NCT02368184
Title: Pilot Study of the CoVa™ Monitoring of Patients With Congestive Heart Failure
Acronym: CoVa
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decided not to go forward with study. No subjects were enrolled.
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-6537
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Congestive Heart Failure
Keywords: noninvasive physiologic monitoring; acute decompensated heart failure (ADHF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to obtain observational data allowing for the preliminary assessment of the utility of a noninvasive physiologic monitor for monitoring of patients with congestive heart failure.

DETAILED DESCRIPTION:
The study proposes to utilize the CoVa™ Monitoring System, a novel body-worn sensor that remotely monitors thoracic fluid, heart rate, heart rate variability, respiration rate, skin temperature, posture, and, using transmitted waveforms, stroke volume and cardiac output to evaluate the system's monitoring capabilities in individuals recently hospitalized for congestive heart failure. The data acquired through this study will play a critical roll in developing future interventional studies that will allow patients with HF to potentially receive better and more timely treatment in the home setting, decreasing hospitalizations and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Have wireless internet access within their homes.
* Acute hospitalization with a primary diagnosis of acute decompensated heart failure (ADHF) diagnosed on the basis of all of the following:

  1. Symptoms:

     * Onset or worsening of dyspnea within the past 2 weeks
  2. Physical exam (at least 1 present):

     * Rales/ Crackles on auscultation
     * Elevated JVP > 8 cmH2O
     * Weight gain
     * LE edema
  3. Diagnostic imaging/ labs (at least 1 present):

     * Evidence of pulmonary congestion or edema on chest X-ray/ chest CT
     * Elevated NT-pro-BNP (age-adjusted) (>1000)
* Patients of particular interest will be those who already have a Medtronic Implantable Cardioverter Defibrillator or Cardiac Resynchronization Therapy device with the OptiVol feature that tracks transthoracic impedance.

Exclusion Criteria:

* Allergy to ECG electrodes
* Psychological or social situation that would make the study difficult for the patient
* Inability to consent
* Pregnant women
* Pneumonia - currently, or within the past 30 days
* Non-cardiogenic pulmonary edema (e.g. ARDS)
* Interstitial lung disease
* End-stage renal disease and on hemodialysis
* For any reason unable to wear or place the CoVa™ device, e.g. pectus excavatum, fragile skin, severe arthritis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be made up of adult men and women admitted to the hospital with a primary clinical diagnosis of acute decompensated heart failure. A convenience sample of 25 individuals meeting the following Inclusion criteria and have no Exclusion criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Track physiologic parameters among patients with ADHF and explore predictive algorithms to allow for early ID of patients at risk of ADHF. | 65 days
  * To track on a daily basis important physiologic parameters among patients with a primary diagnosis of acute decompensated heart failure (ADHF) beginning at the time of their hospitalization and then continued for up to 60 days after discharge, in order to better understand their inter- and intra- individual variability and compare this to standard monitoring including daily weights.
  * To explore the development of predictive algorithms to allow for the early identification of patients at risk of acute decompensation and/or HF hospitalization.

SECONDARY OUTCOMES:
Compare transthoracic impedance in individuals who already have a Medtronic implanted device with OptiVol technology. | 65 days
  Compare transthoracic impedance measured noninvasively with the CoVa and invasively in individuals who already have a Medtronic implanted device with OptiVol technology.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Steinhuble, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No